CLINICAL TRIAL: NCT04367415
Title: Darwish Test (Office Hysteroscopic Bubble Suction and Tubal Peristalsis) in Cases of Intrauterine Polyp(s)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Professor of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Other Study IDs: Darwish test and polyp(s)
Record Dates: First submitted 2020-04-20; First posted 2020-04-29 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Intrauterine Polyp
Keywords: hysteroscopy; tubal patency; bubble suction test; tubal peristalsis; infertility; Abnormal uterine bleeding
MeSH Terms: conditions — Infertility; Metrorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal uterine cavity on office hysteroscopy: If the uterine cavity is normal the patient will be allocated as group A.
  Interventions: Diagnostic Test: Darwish test for a free endometrial cavity; Diagnostic Test: Darwish test for an endometrial cavity with endometrial polyps
- uterine cavity shown one or more polyps on office hysteroscopy: If there is one or more polyp(s) the patient will be allocated as group B. Localization and size estimation of the polyp(s) is mandatory.
  Interventions: Diagnostic Test: Darwish test for a free endometrial cavity; Diagnostic Test: Darwish test for an endometrial cavity with endometrial polyps

INTERVENTIONS:
Diagnostic Test: Darwish test for a free endometrial cavity — Darwish test (Office hysteroscopic bubble suction and tubal peristalsis). If the uterine cavity is normal the patient will be allocated as group A
Diagnostic Test: Darwish test for an endometrial cavity with endometrial polyps — Darwish test (Office hysteroscopic bubble suction and tubal peristalsis).If there is one or more polyp(s) the patient will be allocated as group B.

SUMMARY:
Anatomic Fallopian tubal patency and physiologic patency testing are feasible via hystertoscopy. This study aims to test the impact of different types of intrauterine polyp(s) on Darwish test (office hysteroscopic bubble suction test and tubal peristalsis).

DETAILED DESCRIPTION:
It will include women with suspected intrauterine polyp(s) as diagnosed by transvaginal ultrasonography (TVS) or saline infusion sonography (SIS). They will be women complaining from abnormal uterine bleeding in the form of menorrhagia, metorrhagia, intermenstrual spotting or postcoital bleeding, or infertility. Intrauterine polyp(s) could be included based on a recent hysterosalpingography (HSG) with an intrauterine circumscribed filling defect with sharp border. Preoperative counseling of all patients followed by an informed written consent taken from those who will agree. The included patients subjected to complete history taking and meticulous physical examination. A suspected pregnancy, heavy vaginal bleeding, active pelvic inflammatory disease (PID), severe co-morbidity, e.g., severe cardiac, neurologic, or chest disease, and other medical contraindications to pregnancy will be exclusion criteria of this study. Selected cases will be subjected to office hysteroscopy.

Sample size calculation is based on the investigator's previous study on the prevalence of tubal patency using bubble suction test in infertility patients with normal FT. The percentage of agreement between office hysteroscopy and diagnostic laparoscopy will be 92% and 88% for the right and left tubes respectively. If it is supposed that bubble suction test would be positive in about 90% of apparently normal FT and it would be positive in about 60% of cases with intrauterine polyp(s), sample size in each group would be 51 cases needed to have a confidence level of 95% with α error of 0.05 (the real value is within ±5% of the measured/surveyed value). The vulva, vagina and the thighs will be disinfected with a 10% povidone-iodine solution. Sterile draping will be applied.

Office diagnostic hysteroscopy will be performed using a 2.6 mm 30° rigid scope with a 3.2mm outer sheath (Karl Storz, Tutlingen, Germany). At the beginning in all cases vaginoscopic approach is tried but if any difficulty will be encountered, grasping of the anterior lip of cervix with a volsellum will be done. Therafter, the uterus will be distended with normal saline at 100-150 mmHg generated from a pneumatic cuff of sphygmomanometer wrapped around the 500-cm3 infusion bottle. As attached to a 250-W Xenon light source, the scope will be introduced gently through the cervical canal and internal os. To perfectly perform hysteroscopic tubal patency testing the following tricks should be followed. Clear view of the endometrial cavity should be achieved on panoramic view by placing the hysteroscope at internal os waiting for a while to achieve homogenous distension. The uterine cavity should be systematically examined starting by its anterior and posterior walls, the fundus, and the borders. Examination will be considered complete if the both tubal ostia will be reached describing any gross pathology, e.g., septum, adhesions, polyp(s), myoma, and any growth.

If the uterine cavity is normal the patient will be allocated as group A. If there is one or more polyp(s) the patient will be allocated as group B. Localization and size estimation of the polyp(s) is mandatory.

Prerequisites for a successful access to evaluate tubal patency include utilization of a 300 telescope with gaining skill of its rotation to reach both cornea and most importantly orientation with a fundamental anatomic triad (Darwish triad) (DT). The most proximal corneal fine wide circle is the ostium (the end of the endometrial cavity) representing a base of a cone which is followed by a shallow conical groove (the first millimeters of the intramural part of FT). Finally, a distal pinhole dark spot (the narrowest part of the FT) representing the tip of the cone. Putting DT (ostium, intramural part and dark spot) in mind is the key step to evaluate tubal patency and physiology via hysteroscopy. If DT is clearly accessible, the hysteroscopist should comment on this. If there are some osteal lesions like tiny polyp(s) or fine adhesions that may hinder proper evaluation of the tubal anatomy and physiology, the hysteroscopist should notice and document. Passage of any air bubbles in the irrigating fluid towards DT is reported. If no observed air bubbles, the hysteroscopist should inject just 2 ml of air into the rubber end of the sterile infusion set. Hysteroscopic bubble suction test is considered positive if air bubbles are sucked by DT within 1 min. During this period, neither injection of air nor increased pressure will be done. If no suction of gas bubbles occurred, the examiner should wait for 1 min more to exclude tubal spasm. Again, if no suction of the bubbles by DT and their accumulation at the corneal end, the test will be considered negative. Simultaneously, careful visualization of any change in the shape of the ostium and intramural part of FT particularly during suction of the air bubbles will be recorded in all cases. Tubal peristalsis is defined as observed osteal and intramural tubal rhythmic opening and closing on maintained intrauterine pressure, i.e., periodic changes of DT in the form of widening followed by collapse on meticulous observation. If the ostium and intramural part of the tube is obviously opened followed by collapse and non-visualization of the pinhole dark spot of DT for a while, positive peristalsis will be reported. The same steps will be repeated on the contralateral side and reported.

ELIGIBILITY:
Inclusion Criteria:

* intrauterine polyp(s) as diagnosed by transvaginal ultrasonography (TVS) or saline infusion sonography (SIS).
* abnormal uterine bleeding in the form of menorrhagia, metorrhagia, intermenstrual spotting or postcoital bleeding,
* infertility.

Exclusion Criteria:

* A suspected pregnancy,
* heavy vaginal bleeding,
* active pelvic inflammatory disease (PID),
* severe co-morbidity, e.g., severe cardiac, neurologic, or chest disease, and other medical contraindications to pregnancy

Ages: 20 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: women with suspected intrauterine polyp(s)
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-12-23 (Estimated); Study Completion 2022-12-26 (Estimated)

PRIMARY OUTCOMES:
Anatomic and physiologic tubal patency (Office hysteroscopic bubble suction and tubal peristalsis) in cases of intrauterine polyp(s) | 1 year
  diagnostic test

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided